CLINICAL TRIAL: NCT05339893
Title: Evaluating the Use of Trans Auricular Vagus Nerve Stimulation (taVNS) and Robotic Training to Improve Upper Limb Motor Recovery After Stroke
Brief Title: Trans Auricular Vagus Nerve Stimulation (taVNS) and Robotic Training for Paralyzed Arm After Stroke
Acronym: VaNSaRTS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Professor, Investigator, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-1355
Record Dates: First submitted 2022-03-29; First posted 2022-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Hemiparesis
Keywords: taVNS; Trans Auricular Vagus Nerve Stimulation; Robotic Training; Upper Limb Motor Recovery
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Intervention Model Description: To determine whether treatment with taVNS during the robotic training of a patient with stroke and a paralyzed arm will alter the motor impairment.
Who Masked: Participant, Investigator
Masking Description: The patient will not know whether they are receiving taVNS, all patients will feel a tingling in the ear as the current is ramped up and then down to determine a stimulation threshold, but only the active group will receive timed stimulation bursts during the robotic protocol that engages the affected limb. The measuring clinician will not know a patient's group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Affected Limb (Sham Comparator): Patients will wear the taVNS device on the left ear for the duration of the subsequent phase of the robotic training. During this phase the patient will engage the robotic device with the affected limb and complete the protocol and the stimulation or sham stimulation will occur with every extensor movement.
  Within subject. Sham controlled. Double blind, the patient will not know whether they are receiving taVNS, all patients feel a ramp up current but only the active group will receive timed stimulation bursts during the robotic protocol that engages the affected limb. '
  Interventions: Device: In Motion Rehabilitation Robot
- Unaffected limb (No Intervention): Patients will engage the robot first with their unaffected limb. This practice will ensure understanding and serve to activate the hemisphere ipsilateral to the impaired limb. Patients are likely to perform this activity quickly, there will not be any taVNS during this part of the procedure.

INTERVENTIONS:
Device: In Motion Rehabilitation Robot — Patients will wear the taVNS device on the left ear for the duration of the subsequent phase of the robotic training. During this phase the patient will engage the robotic device with the affected limb and complete the protocol and the stimulation or sham stimulation will occur with every extensor movement.
  Arms: Affected Limb

SUMMARY:
To determine whether treatment with transauricular vagus nerve stimulation (taVNS) during the training of an affected upper limb of a patient with chronic stroke on a robotic motor task alters the motor impairment.

DETAILED DESCRIPTION:
The investigators will evaluate whether transauricular vagus nerve stimulation (taVNS) delivered during extensor movements executed on a robotic device will alter the clinical measurement of upper limb motor performance in 45 patients with chronic stroke.

Patients will engage the robot first with their unaffected limb. This practice will ensure understanding and serve to activate the hemisphere ipsilateral to the impaired limb. Patients are likely to perform this activity quickly, there will not be any taVNS during this part of the procedure. Patients will then wear the taVNS device on the left ear for the duration of the subsequent phase of the robotic training. During this phase the patient will engage the robotic device with the affected limb and complete the protocol and the stimulation or sham stimulation will occur with every extensor movement.

ELIGIBILITY:
Inclusion Criteria:

* In receipt of full vaccination status and no recent upper respiratory symptoms and no loss of taste or olfaction.
* Individuals between 18 and 85 years of age
* First single focal unilateral supratentorial ischemic stroke with diagnosis verified by brain imaging (MRI or CT scans) that occurred at least 6 months prior
* Cognitive function sufficient to understand the experiments and follow instructions (per interview with Speech Pathologist or PI)
* Fugl-Meyer assessment 12 to 44 out of 66 (neither hemiplegic nor fully recovered motor function in the muscles of the shoulder, elbow, and wrist).

Exclusion Criteria:

* Recent fever or upper respiratory symptoms.
* Botox treatment within 3 months of enrollment
* Fixed contraction deformity in the affected limb
* Complete and total flaccid paralysis of all shoulder and elbow motor performance
* Prior injury to the vagus nerve
* Severe dysphagia
* Introduction of any new rehabilitation interventions during study
* Individuals with scar tissue, broken skin, or irremovable metal piercings that may interfere with the stimulation or the stimulation device
* Highly conductive metal in any part of the body, including metal injury to the eye; this will be reviewed on a case by case basis for PI to make a determination
* Pregnant or plan on becoming pregnant or breastfeeding during the study period
* Significant arrhythmias, including but not limited to, atrial fibrillation, atrial flutter, sick sinus syndrome, and A-V blocks (enrollment to be determined by PI review)
* Presence of an electrically, magnetically or mechanically activated implant (including cardiac pacemaker), an intracerebral vascular clip, or any other electrically sensitive support system; Loop recorders will be reviewed on a case by case basis by PI and the treating Cardiologist to make a determination

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2024-04-18 (Estimated); Study Completion 2025-04-18 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Scale for the upper extremity | 30-45minutes
  A standard well characterized measure of the movement ability of the subjects arm- shoulder, elbow, wrist, hand and fingers.

SECONDARY OUTCOMES:
Action Research Arm Test (ARAT) | 30-45minutes
  A standard evaluation of 19 different real world actions of the arm, including movements around the shoulder, elbow, wrist, hand and fingers.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce T Volpe, MD, Principal Investigator — Feinstein Center for Molecular Medicine; Timir Datta Chaudhuri, PhD, Study Director — Feinstein Center for Bioelectronic Medicine
Locations (1):
- Feinstein Institutes at Northwell Health, Manhasset, New York, United States